CLINICAL TRIAL: NCT04513535
Title: A Comparison of the Effects of Cervical and Thoracic Manipulation, Glenohumeral Mobilization, and Sleeper Stretch on Shoulder Strength and Range of Motion in Healthy Individuals
Brief Title: Effects of Manual Therapy on Shoulder Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PRO20010001
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Musculoskeletal Manipulations; Shoulder; Range of Motion; Muscle Strength; Surface Electromyography
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: modified crossover, each group will experience 2/4 interventions
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor blinded to group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- manual therapy combination 1 (Experimental): Cervical manipulation, Thoracic manipulation
  Interventions: Other: Thoracic Manipulation; Other: Cervical Manipulation
- manual therapy combination 2 (Experimental): Cervical manipulation, glenohumeral mobilization
  Interventions: Other: Cervical Manipulation; Other: glenohumeral posterior glide mobilization
- manual therapy combination 3 (Experimental): cervical manipulation, sleeper stretch
  Interventions: Other: Cervical Manipulation; Other: Sleeper stretch
- manual therapy combination 4 (Experimental): thoracic manipulation, glenohumeral mobilization
  Interventions: Other: Thoracic Manipulation; Other: glenohumeral posterior glide mobilization
- manual therapy combination 5 (Experimental): thoracic manipulation, sleeper stretch
  Interventions: Other: Thoracic Manipulation; Other: Sleeper stretch
- manual therapy combination 6 (Experimental): glenohumeral mobilization, sleeper stretch
  Interventions: Other: glenohumeral posterior glide mobilization; Other: Sleeper stretch

INTERVENTIONS:
Other: Thoracic Manipulation — A supine thoracic manipulation will be utilized. Participants will be lying supine on the plinth with their arms crossed over their chest, making sure the forearms are not crossed. An experienced clinician will place their hand on the inferior segment (T4); the superior segment (T3) will be placed in the midrange of thoracic flexion and extension. The clinician will apply a high velocity, end range, anterior to posterior thrust by using their body weight to deliver the thrust through the participants crossed elbows, thus creating a bilateral gapping of the facet joints. If a cavitation is achieved after the first thrust, the thoracic manipulation intervention is complete. If not, one more attempt will be made to achieve a cavitation. Regardless of if there was a cavitation or not, after the second attempt the intervention is complete.
  Arms: manual therapy combination 1; manual therapy combination 4; manual therapy combination 5
Other: Cervical Manipulation — Participants will be lying supine on the plinth on the table. A high velocity low amplitude manipulation will be performed to the cervical spine by an experienced clinician.The clinician will place the right proximal phalanx of the index finger over the posterolateral aspect of the articular pillar at the right C4/C5 segment to maximally influence the C5 myotomal distribution. The clinician's left hand will be cradling the participants head. The participant will be brought into midrange flexion-extension, ipsilateral side bend, and contralateral rotation of C4/5. Once a firm end feel is felt the manipulation will be administered into left rotation in an arc toward the left eye. If a cavitation is achieved after the first thrust, the intervention is complete. If not, one more attempt will be made to achieve a cavitation;after the second attempt the intervention is complete.
  Arms: manual therapy combination 1; manual therapy combination 2; manual therapy combination 3
Other: glenohumeral posterior glide mobilization — Participants will be instructed to lay supine on the plinth and a plastic orthopedic wedge will be placed under their scapula for stabilization on the side that is receiving the mobilization. The experienced clinician will stand on the same side being mobilized and held the participant's arm proximal to the medial and lateral humeral epicondyles. The clinician will hold the participant's arm in the scapular plane, approximately 55 degrees of abduction and slight ER with a grade one long axis distraction applied and sustained throughout the entire mobilization. A grade three oscillatory mobilization will be applied for three sets of 30 seconds with a 30 second rest in between.
  Arms: manual therapy combination 2; manual therapy combination 4; manual therapy combination 6
Other: Sleeper stretch — Participants will be positioned in a side lying position with the arm to be stretched on the table. The arm to be tested will then be positioned at a 90-90 shoulder abduction and elbow flexion position. A support will be positioned behind the patient to ensure there is no compensatory trunk movement during the stretch, and an examiner verified the arm is in a 90-90 position. A sleeper stretch will be subsequently completed, in which the participant will internally rotate the arm to stretch the posterior shoulder musculature. Three, thirty second stretches will be completed
  Arms: manual therapy combination 3; manual therapy combination 5; manual therapy combination 6

SUMMARY:
The purpose of this study is to directly compare the effects of four distinct interventions commonly used in the treatment of shoulder pathology on shoulder range of motion (ROM) and strength in asymptomatic shoulders:

* grade III oscillatory anterior-posterior glenohumeral joint mobilizations
* an internal rotation (IR) "sleeper" stretch
* supine upper-thoracic manipulation
* cervical spine manipulation

DETAILED DESCRIPTION:
Research questions:

Do different interventions result in different immediate changes in shoulder ROM? Ha1: Stretching and glenohumeral mobilization will result in increased shoulder ROM Ha2: Thoracic and Cervical manipulations will result in decreased shoulder ROM Ho: There will be no differences in shoulder ROM between groups for each of the four interventions

Do different interventions result in different immediate effects for shoulder external rotation (ER) strength? Ha1: Stretching and glenohumeral mobilization will result in a decrease in ER strength Ha2: Thoracic and cervical manipulations will result in increased ER strength Ho: There will be no differences in ER strength between groups for each of the four interventions

Do different interventions result in different immediate effects for shoulder electromyographic (EMG) activity? Ha1: Stretching and glenohumeral mobilization will result in a decrease in EMG activity Ha2: Thoracic and cervical manipulations will result in increased EMG activity Ho: There will be no differences EMG activity between groups for each of the four interventions

Based on pilot data, the apparent effect sizes ranged from .57 - .78. With the ɑ = .05 and 1-β = .80, G-power software for a 4 group ANOVA yields a sample of 20 participants per group. To account for possible sample variations and participant drop-outs, a sample of 24 per group will be enrolled. Based on the study design of a randomized cross-over study, where each participant will receive two of the interventions, a total sample of 48 individuals will be enrolled.

Once a participant is cleared to participate, all individuals will undergo the following tests:

External Rotator Strength Test Strength of the external rotators (infraspinatus) will be measured by a blinded examiner using a hand-held dynamometer (Micro-FET 2, Hoggan Health Industries, Salt Lake CIty, UT). The dynamometer will be placed on the high threshold setting and the force recorded in Newtons. The strength measurement will be taken with the participant in the prone position with their shoulder abducted 90 degrees and 80 degrees of external rotation with the elbow bent to 90 degrees. Abduction (ABD) and elbow flexion ROM positioning will be assessed using a goniometer, and the shoulder external rotation ROM will be measured using the iPhoneX. To ensure consistent placement, the researchers will place a mark 10 cm proximal to the medial epicondyle of the humerus. This mark will be aligned with the edge of the table in order to allow for adequate clearing of the arm and dynamometer while completing the test. A second mark will be placed on the distal end of the radius, using the radial styloid process as a reference. The distal edge of the dynamometer will be placed at this mark. The testers knee will be positioned behind the participant's elbow to ensure there is no compensation and activation of other muscles. At the start of the test the participant will be instructed to resist the pressure applied by the tester. The tester will apply their force progressively over 5 seconds while the participant maximally resists against the dynamometer plate. Two pretest and two post-test measurements of strength will be obtained, with the greater measurement used for data analysis.

Posterior Shoulder Tightness Posterior shoulder tightness (PST) will be measured by blinded examiners with the participant side lying with hips and knees flexed to 45 degrees. The non-tested humerus will be placed behind the participants head with half of their humerus off of the plinth. The participants' arm being tested will be placed so that the humeral condyles will be stacked perpendicular to the plinth with the olecranon facing posteriorly in relation to the participants' body. The participant's arm will be marked 5cm proximal to the lateral epicondyle, where an independent examiner will place the top of the iPhoneX to measure PST in degrees. The Level in the Measure application, manufactured by Apple's arkit via iOS 13.2.3, will be used to measure horizontal adduction and quantify PST. The tester will be blinded from the results of the PST measurement. The arm being tested will be gripped by the tester just distal to the humeral condyles. The scapula will be stabilized in retraction throughout the test. The test will be completed and the measurement will be recorded when the tester is no longer able to stabilize the scapula or the movement ceases. Two trials will be performed by the tester with a 10 second rest between trials.

Internal Rotation ROM Internal rotation range of motion will be measured by a blinded examiner with the participant in the prone position, shoulder abducted to 90 degrees, with a bolster under the mid-humerus to keep the glenohumeral joint in the neutral position. A mark will be placed on the participants arm 5cm distal to the medial epicondyle on the ventral forearm where the top of the iPhoneX will be placed to measure internal rotation range of motion in degrees. Two testers will be used to complete the test. One tester will apply stabilization by placing their elbow atop the scapula, their forearm on top of the participant's humerus, and take the participants through the motion. The other tester will hold the iPhoneX and record the final measurement. The test will be completed when the scapula begins to rise from the table or no further motion is felt. The tester performing the motion will be blinded to the measurements being taken. Two trials will be taken on the right upper extremity.

The iPhoneX (iOS 13.2.3) will be used as an inclinometer using the Level in the Measure application that is pre-downloaded on the iPhoneX. In this study, the smartphone inclinometer application that is available to iPhones for purchase was used.

EMG of the Infraspinatus Pre-post intervention activity of the infraspinatus muscle will be assessed with surface EMG during a maximal voluntary isometric contraction (MVIC). Before placing the electrodes on the participants, the area will be thoroughly cleaned with an alcohol wipe. A single, Norotrode 20 electrode will then be placed over the muscle belly of the infraspinatus. The Delsys EMGworks acquisition software will be used to obtain all EMG data. The electrodes will be sampled at a rate of 1926 samples/s. Maximal Voluntary Isometric Contraction (MVIC) will be recorded simultaneously with the isometric strength testing. The MVC for each participant consists of a 5s hold in the standard manual muscle testing(MMT) positioning.

All EMG data will be prepared and collected by an assessor blinded to the assigned intervention, and will be analyzed using the Delsys EMGworks Analysis software.

Randomization:

Prior to enrollment, using paired, block randomization, a set of 48 group assignments will be prepared and placed in sealed, opaque envelopes by an individual not involved in the data collection process.

The participants will be assigned to two of the four different intervention groups: posterior shoulder mobilization, cervical manipulation, thoracic manipulation, and a self-applied sleeper stretch technique.

All participants will select an envelope at the time of enrollment, and only reveal the contents to the examiner preforming the intervention. The first intervention will be applied at the first research session, and the second intervention will be applied during a second session approximately one week later.

Data Analysis:

Baseline and participant demographic data will be analyzed and reported using descriptive and measures of central tendency.

Interaction and main effects for Internal rotation ROM, posterior shoulder tightness, external rotation force, and infraspinatus EMG activity x intervention will be assessed with repeated measures ANOVAs and post hoc testing.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in this study if they:

  * are between the ages of 18 and 55
  * have no history of shoulder, neck, or upper back dysfunction.

Exclusion Criteria:

* Individuals will be excluded if they report having any of the following conditions:

  * shoulder, neck, or upper back pain;
  * prior shoulder, neck or upper back surgery;
  * previous injury to shoulder, neck, or thoracic area;
  * active inflammatory disease process in treatment area;
  * osteoporosis;
  * signs and symptoms of a nerve root pathology/radiculopathy (dermatomal sensory changes, myotomal weakness, reflex changes);
  * upper motor neuron lesions/spinal cord pathology;
  * local infection;
  * active or history of cancer;
  * long term corticosteroid use;
  * systemically unwell;
  * systemic hyperlaxity;
  * known connective tissue disease;
  * known abnormalities of the spine;
  * disturbance of bowel or bladder;
  * coronary artery disease;
  * unstable upper cervical spine;
  * positive testing for vertebral basilar insufficiency (VBI);
  * spondylolisthesis;
  * spondylosis;
  * pregnancy or recent pregnancy;
  * nervous system dysfunction;
  * has received physical therapy for related shoulder, neck, or upper thoracic dysfunction;
  * blood clotting disorder;
  * receiving workman's compensation or involved in an active lawsuit;
  * currently taking fluoroquinolones (Cipro, Factive, Levaquin, Avelox, Noroxin, Floxin)
  * any other known contraindication to manual therapy The study will not include adults unable to consent/persons with cognitive/developmental disability, individuals who are not yet adults, pregnant women, or prisoners or other detained individuals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in shoulder ER strength | immediate pre-post intervention
  pre-test post-test strength test of the infraspinatus with hand held dynamometer
Change in shoulder IR ROM | immediate pre-post intervention
  change pre-post test IR ROM at 90 degrees ABD
change in posterior shoulder mobility | immediate pre-post intervention
  change in pre-post test posterior shoulder mobility assessed in horizontal adduction
change in infraspinatus EMG activity | immediate pre-post intervention
  change in pre-post test EMG peak and mean root squared activity

CONTACTS AND LOCATIONS:
Overall Officials: Brian Swanson, PT, DSc, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be made available in de-identified form upon request